CLINICAL TRIAL: NCT04865731
Title: A Phase II Clinical Trial of Dermaprazole Cream for Radiation Dermatitis in Head and Neck Cancer Patients (CTMS# 20-0147)
Brief Title: Dermaprazole Cream for Radiation Dermatitis in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTMS# 20-0147; HSC20210301H (Other: UT Health San Antonio)
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Cancer of the Head and Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Esomeprazole; Petrolatum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dermaprazole (Experimental): 30 HNC patients who will be using Dermaprazole twice daily for 7 weeks
  Interventions: Drug: Dermaprazole
- Aquaphor (Active Comparator): 15 HNC patients using Aquaphor, the current clinical standard of care
  Interventions: Drug: Aquaphor

INTERVENTIONS:
Drug: Dermaprazole — Patients will be managed with twice daily prophylactic use of the proposed intervention (Dermaprazole) topical cream for radiation dermatitis. The amount of cream will be 2cc per application and will be measured in pre-filled capped syringes for every application.
  Other Names: esomeprazole
  Arms: Dermaprazole
Drug: Aquaphor — Patients will be managed with twice daily prophylactic use of Aquaphor. The amount of Aquaphor will be 2cc per application and will be measured in pre-filled capped syringes for every application.
  Arms: Aquaphor

SUMMARY:
In this study, the study team seek to conduct a pilot clinical study to evaluate the safety and efficacy of a reformulated proton pump inhibitor (PPI) cream (Dermaprazole) in definitive head and neck cancer (HNC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck malignancy (including radiation therapy to primary head cancers of any histology and/or neck lymphatics, excluding brain malignancies)
* Biopsy proven diagnosis of head and neck malignancy
* Planned to receive definitive chemoradiation of at least 66Gy
* Age 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Written Informed Consent
* History and Physical within 12 weeks of enrollment

Exclusion Criteria:

* Prior head and neck radiotherapy
* Neoadjuvant chemotherapy
* Any serious medical condition or illness that would preclude the safe administration of the trial treatment including, but not limited to, active infection, symptomatic heart failure, unstable angina, psychiatric illness or social situations that would limit compliance with treatment
* Currently taking proton pump inhibitors. Eligible if discontinues with physician approval.
* Lack of concurrent chemotherapy
* Open wound at time of simulation
* Known autoimmune, connective tissue, or skin disorder; or other theoretical radiosensitivity to include bullous pemphigoid, dermatomyositis, lupus of the skin and scleroderma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shraddha Dalwadi, MD, Principal Investigator — The University of Texas Health Science Center - Mays Cancer Center
Locations (1):
- Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Dermaprazole: HNC patients who will be using Dermaprazole twice daily for 7 weeks
  Dermaprazole: Patients will be managed with twice daily prophylactic use of the proposed intervention (Dermaprazole) topical cream for radiation dermatitis. The amount of cream will be 2cc per application and will be measured in pre-filled capped syringes for every application.
- Aquaphor: HNC patients using Aquaphor, the current clinical standard of care
  Aquaphor: Patients will be managed with twice daily prophylactic use of Aquaphor. The amount of Aquaphor will be 2cc per application and will be measured in pre-filled capped syringes for every application.
Period: Overall Study
Arm/Group | Dermaprazole | Aquaphor
Started | 4 | 2
Completed | 1 | 0
Not Completed | 3 | 2
Not completed — Physician Decision | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants receiving radiation therapy
Groups:
- Total: Total of all reporting groups
Arm/Group | Dermaprazole | Aquaphor | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Rates of Clinically Significant Radiation Dermatitis as Defined as NCI CTCAE Version 5 Grade 2 or Higher
Description: Number of radiation dermatitis adverse events defined by the NCI CTCAE version 5 that are graded as 2 or higher
Time Frame: 15 months
Measure: Number; unit: Number of events
Arm/Group | Dermaprazole | Aquaphor
Number analyzed (Participants) | 4 | 2
Number of events | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline to 15 months
Description: Adverse events considered to be possible or probably or definitely related to intervention. For purposes of this study, an adverse event is considered expected when the events are those related to systems within the radiation treatment field and include: infection, allergy, or short & long-term (greater than 6 month) skin changes.
Arm/Group | Dermaprazole | Aquaphor
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dermaprazole (N=4) | Aquaphor (N=2)
Anemia (Blood and lymphatic system disorders) | 2 (3) | 1 (5)
Anorexia (Gastrointestinal disorders) | 1 (8) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (3) | 0 (0)
Dermatitis radiation (Skin and subcutaneous tissue disorders) | 4 (11) | 2 (5)
Anosmia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (21) | 2 (5)
Dysgeusia (Gastrointestinal disorders) | 4 (14) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 3 (18) | 1 (1)
Ear and Labyrinth disorders (Ear and labyrinth disorders) | 2 (6) | 0 (0)
Fatigue (General disorders) | 4 (10) | 1 (3)
Hoarsness (General disorders) | 2 (2) | 0 (0)
Lymphedema (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (12) | 2 (8)
Myelitis (Immune system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (15) | 2 (5)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Oropharyngeal pain (Gastrointestinal disorders) | 1 (5) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (16) | 1 (1)
Trismus (Gastrointestinal disorders) | 0 (0) | 1 (5)
Vomiting (Gastrointestinal disorders) | 1 (4) | 0 (0)
Weight loss (Gastrointestinal disorders) | 3 (15) | 1 (3)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 1 (4)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypercalcemia (General disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
White Blood Cell decrease (Blood and lymphatic system disorders) | 2 (8) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04865731/Prot_SAP_000.pdf